CLINICAL TRIAL: NCT01998321
Title: Bilateral Simultaneous Total Knee Arthroplasty in Patients With Severe Articular Deformities
Brief Title: PSI for Bilateral Simultaneous TKA in Sever Varus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: October 6 University (Other)
Responsible Party: Principal Investigator, Mahmoud A Hafez, MSc Orth, Dip SICOT, FRCS Ed, MD, Mahmoud A Hafez, October 6 University
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: October6U-0002
Record Dates: First submitted 2013-11-16; First posted 2013-11-28 (Estimated); Last update posted 2013-11-28 (Estimated); Status verified 2013-11

CONDITIONS: Knee Osteoarthritis
Keywords: PSI: Patient Specific Instrument; TKA: Total Knee Arthroplasty; Articular Deformity; Varus
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TKA using PSI (Experimental): Total Knee Arthroplasty using Patient Specific Instrument
  Interventions: Other: Patient specific instrument
- 2 TKA using conditional technique. (Experimental): Total Knee Arthroplasty using conditional technique.
  Interventions: Other: conventional technique for TKA

INTERVENTIONS:
Other: Patient specific instrument — A special software with the ability to perform 3D planning including sizing, alignment, bone cutting, positioning of implants, simulation & PSI designing and PSI production
  Other Names: PSI
  Arms: TKA using PSI
Other: conventional technique for TKA
  Arms: 2 TKA using conditional technique.

SUMMARY:
the Purpose of this study was to evaluate the short term outcome of patient specific instrument (PSI) in cases of bilateral simultaneous total knee arthroplasty (TKA) for knee osteoarthritis with sever varus

DETAILED DESCRIPTION:
The incidence of knee Osteoarthritis is variable and it is very high in Far East 47.0% and 70.2% in men and women respectively, while it is 17.2% and 82.8% in male and females respectively in Middle East. The incidence of bilateral knee Osteoarthritis is 48%. TKA is the standard treatment for Osteoarthritis. Many authors prefer bilateral simultaneous TKA can be performed for straight forward cases of Knee Osteoarthritis, although it has higher complication rate that could be discouraging.

Knee Osteoarthritis could be associated with articular deformities such as varus, valgus, flexion deformity and rarely recurvatum. These deformities could be associated with bone loss, ligamentous laxity, leg length discrepancy, bilateral shortening and disfigurement. These deformities need to be corrected during TKA and this make the procedure more difficult especially in severe cases with associated problems as described above. Some patients with knee Osteoarthritis present late when the condition becomes bilateral with sever articular deformity. Late presentation is a common feather in developing countries and low income countries and also in Middle and Far East.

With the progression of Knee Osteoarthritis patient's condition deteriorates gradually, both local and generally with increasing loss of cartilage and bone leading to deformities and joint laxity. This general condition with the increasing disability leads to high risk of associated obesity and comorbidities. The late presentation is multifactorial and complex to explain. There are obvious reasons such as economic constrain, late referral, lake of experienced surgeons and high demand and expectation such as full flexion in Middle and Far East. There are other unexplained reasons such as fear of surgeries, misconception about TKA and psychological factors.

Unilateral TKA for patients with bilateral knee Osteoarthritis with sever articular deformities is not beneficial to the patients, as it does not allow correction of the deformities and easier rehabilitation, and may not be satisfying for the patient because patient left with a straight knee after TKA and a deformed knee in the other side that leads to difficult rehabilitation and may force the TKA to get the same deformity to adapt to the other knee. With this dissatisfaction the patient may refuse to have the other knee done.

Bilateral simultaneous TKA in patient with sever articular deformities is beneficial to the patients as it allows correction of the deformities and easier rehabilitation.

However bilateral simultaneous TKA for such complex cases is a very demanding procedure and could be associated with a higher rate of complications such as fat embolism , mortality, infection, bleeding, deep venous thrombosis, and general complications.

PSI could be useful for bilateral simultaneous TKA because it eliminates the use of intramedullary guides and may reduce operative time, bleeding and risk of complications such as fat embolism or infection.

The aim of this study is to review the outcome of using PSI in bilateral simultaneous TKA for patient with sever articular deformities which is common in middle east region.

ELIGIBILITY:
Inclusion Criteria:

* Deformity ranging from 5 to 30 varus,
* 10-40 valgus,
* fixed flexion deformity from 5 to 50
* wellness to participate in the study

Exclusion Criteria:

* absence of deformities varus, valgus, or flexion deformity

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2012-12; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
functional score | up to 52 weeks

SECONDARY OUTCOMES:
Blood transfusion rate | up to 52 weeks
complication rate | up to 52 weeks
hospital stay | up to 52 weeks
Operative time | during surgery

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud A Hafez, Professor, Principal Investigator — October 6 University; Mohamed El Sayed, Dr, Study Chair — Bone and Joint Center
Locations (1):
- October 6 University, October Six City, Egypt